CLINICAL TRIAL: NCT04928742
Title: Online Public Health Nurse-Delivered Group Cognitive Behavioural Therapy for Postpartum Depression
Brief Title: Online PHN CBT for PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, MD, PhD, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OnlinePHNCBT
Record Dates: First submitted 2021-04-09; First posted 2021-06-16 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to the treatment group (online PHN-delivered group CBT) or the control group (treatment as usual).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator, outcome assessors and data analysts will be blinded to participant allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (9-week online CBT group) (Experimental): Participants assigned to the treatment group will participate in a 9-week group CBT intervention for PPD delivered via Zoom by two public health nurses. This intervention was developed by Dr. Van Lieshout (PI) at the Women's Health Concerns Clinic (WHCC) at St. Joseph's Healthcare Hamilton. It was designed to be brief, simple, and applicable to women in community settings. It consists of 9 weekly 2-hour sessions where core CBT skills are learned and practiced, and a new psychoeducational topic is introduced and discussed by women each week. All participants in the treatment group will be mailed a hardcopy of the program manual.
  Interventions: Behavioral: Group Cognitive Behavioural Therapy (CBT)
- Control (treatment as usual) (No Intervention): The control group will receive standard postnatal care from Niagara Region Public Health, their obstetrician, midwife, and/or family physician.

INTERVENTIONS:
Behavioral: Group Cognitive Behavioural Therapy (CBT) — The 9-week group CBT intervention for PPD delivered via Zoom by two public health nurses. This intervention was developed by Dr. Van Lieshout (PI) at the Women's Health Concerns Clinic (WHCC) at St. Joseph's Healthcare Hamilton. It was designed to be brief, simple, and applicable to women in community settings. It consists of 9 weekly 2-hour sessions where core CBT skills are learned and practiced, and a new psychoeducational topic is introduced and discussed by women each week.
  Arms: Treatment (9-week online CBT group)

SUMMARY:
The primary objective of this study is to determine if online group CBT for PPD delivered by public health nurses is superior to postnatal care as usual in: a) acutely treating PPD, b) reducing relapse and recurrence, c) improving common comorbidities and complications of PPD including anxiety and the mother-infant relationship, and d) to determine if this treatment is cost-effective.

DETAILED DESCRIPTION:
A prospective, 1-site, parallel group, RCT (1:1 ratio) in which outcome assessors and data analysts will be blinded to maternal treatment will be used to compare online PHN-delivered group CBT for PPD to postnatal care as usual.

The primary objective of this study is to determine if online group CBT for PPD delivered by public health nurses is superior to postnatal care as usual in: a) acutely treating PPD, b) reducing relapse and recurrence, c) improving common comorbidities and complications of PPD including anxiety and the mother-infant relationship, and d) to determine if this treatment is cost-effective.

Women in the treatment group will participate in a 9-week group CBT intervention for PPD delivered via Zoom by two public health nurses. It consists of 9 weekly 2-hour sessions where core CBT skills are learned and practiced, and a new psychoeducational topic is introduced and discussed by women each week.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women will be >18 years of age, understand and speak English (so that they can participate in the CBT group and complete study measures), have an EPDS score between of 10 or more and meet diagnostic criteria for current major depressive disorder on the Mini International Neuropsychiatric Interview-Plus (MINI-Plus). They will also all be within 12 months of delivering an infant.

Exclusion Criteria:

* In order to increase the relevance and generalizability of our findings, women can have psychiatric comorbidities with the exception of bipolar disorder, a current psychotic, substance or alcohol use disorder, or antisocial or borderline personality disorder. These are predictors of significant difficulty participating in therapy groups and/or non-response to CBT.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Maternal Depressive Symptoms | 9 weeks
  Edinburgh Postnatal Depression Scale (EPDS): The EPDS is the 10-item gold standard measure of maternal depressive symptoms. A score >12 is consistent with PPD and changes in scores of 4 or more points are indicative of clinically significant improvement.

SECONDARY OUTCOMES:
Anxiety | 9 weeks
  Penn State Worry Questionnaire (PSWQ): The PSWQ is a 16-item self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD.
Mother-Infant Bonding | 9 weeks
  Postpartum Bonding Questionnaire: The Postpartum Bonding Questionnaire is a 25 item maternal report scale that is designed to detect disorders of the mother-infant relationship on four subscales: bonding, rejection and anger, infant-focused anxiety, and incipient abuse.
Social Support | 9 weeks
  The Social Provisions Scale: The SPS is a 24-item self-report measures of the degree to which an individual's social relationships provide support.
Social Support | 6 months
  The Social Provisions Scale: The SPS is a 24-item self-report measures of the degree to which an individual's social relationships provide support.
Relationship with Partner | 6 months
  Dyadic Adjustment Scale: a 32 item scale that assesses partner relationship on 4 subscales: dyadic consensus, affectional expression, dyadic satisfaction and dyadic cohesion.
Relationship with Partner | 9 weeks
  Dyadic Adjustment Scale: a 32 item scale that assesses partner relationship on 4 subscales: dyadic consensus, affectional expression, dyadic satisfaction and dyadic cohesion.
Infant Temperament | 9 weeks
  Infant Behavior Questionnaire-Revised (very short form): Temperament refers to the ways individuals think, behave, and react and is heavily influenced by the degree to which infants and toddlers can regulate their emotions. Factor analysis of the domains of temperament assessed by the IBQ-R (VSF) indicates that they are consistent with 3 broad dimensions of temperament: emotion regulation, negative affectivity, and extraversion. These subscales have demonstrated good internal consistency and inter-rater reliability between parents. Mothers and fathers will complete the IBQ-R on their infants immediately before treatment, right after treatment, and at 6 months afterward.
Infant Temperament | 6 months
  Infant Behavior Questionnaire-Revised (very short form): Temperament refers to the ways individuals think, behave, and react and is heavily influenced by the degree to which infants and toddlers can regulate their emotions. Factor analysis of the domains of temperament assessed by the IBQ-R (VSF) indicates that they are consistent with 3 broad dimensions of temperament: emotion regulation, negative affectivity, and extraversion. These subscales have demonstrated good internal consistency and inter-rater reliability between parents. Mothers and fathers will complete the IBQ-R on their infants immediately before treatment, right after treatment, and at 6 months afterward.
Cost Effectiveness - costs | 9 weeks
  Cost-effectiveness will be measured using incremental cost per quality-adjusted life year ratio.
  Costs: Canadian Community Health Survey and the Service Use and Resources Form. We will measure resources consumed over the trial period from the perspective of public health care payer. Corresponding unit costs will be calculated using provincial or other standard billing rates.
Cost Effectiveness - QALY | 9 weeks
  Cost-effectiveness will be measured using incremental cost per quality-adjusted life year ratio.
  Quality-Adjusted Life Year (QALY): The EQ-5D-5L is a utility-based health-related quality of life instrument consisting of five questions covering depression/anxiety, usual activities, self-care, pain/ discomfort, and mobility. Its validity in measuring the impact of depression is established. Its Canadian scoring algorithm will be used to convert the five responses to health utility at each measurement occasion.
Cost Effectiveness - costs | 6 months
  Cost-effectiveness will be measured using incremental cost per quality-adjusted life year ratio.
  Costs: Healthcare resource utilization data will be collected using a questionnaire based on the Canadian Community Health Survey and the Service Use and Resources Form. We will measure resources consumed over the trial period from the perspective of public health care payer. Corresponding unit costs will be calculated using provincial or other standard billing rates.
Cost Effectiveness - QALY | 6 months
  Cost-effectiveness will be measured using incremental cost per quality-adjusted life year ratio.
  Quality-Adjusted Life Year (QALY): The EQ-5D-5L is a utility-based health-related quality of life instrument consisting of five questions covering depression/anxiety, usual activities, self-care, pain/ discomfort, and mobility. Its validity in measuring the impact of depression is established. Its Canadian scoring algorithm will be used to convert the five responses to health utility at each measurement occasion.
Maternal Major Depressive Disorder | 6 months
  Mini International Neuropsychiatric Interview (MINI): The MINI is a validated structured diagnostic interview used to assess psychiatric disorders consistent with the DSM-IV. It demonstrates very good agreement with the Structured Clinical Interview for DSM-IV and strong inter-rater reliability has been noted.
  Major Depressive Disorder Module: Our primary outcome (recurrence) will be assessed at 6 months post-treatment, but in order to compare trajectories of recovery/recurrence/relapse, we will assess these outcomes at baseline, 9 weeks, and 6 months. Relapse will be assessed at 6 months post-CBT completion.
  Our primary outcome for maternal depression using the MINI will be the proportion of women who meet MINI current MDD diagnostic criteria at 6 months.
Anxiety | 6 months
  Penn State Worry Questionnaire (PSWQ): The PSWQ is a 16-item self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD.
Mother-Infant Bonding | 6 months
  Postpartum Bonding Questionnaire: The Postpartum Bonding Questionnaire is a 25 item maternal report scale that is designed to detect disorders of the mother-infant relationship on four subscales: bonding, rejection and anger, infant-focused anxiety, and incipient abuse.
Maternal Major Depressive Disorder | 9 weeks
  Mini International Neuropsychiatric Interview (MINI): The MINI is a validated structured diagnostic interview used to assess psychiatric disorders consistent with the DSM-IV. It demonstrates very good agreement with the Structured Clinical Interview for DSM-IV and strong inter-rater reliability has been noted.
  Major Depressive Disorder Module: Our primary outcome (recurrence) will be assessed at 6 months post-treatment, but in order to compare trajectories of recovery/recurrence/relapse, we will assess these outcomes at baseline, 9 weeks, and 6 months. Relapse will be assessed at 6 months post-CBT completion.
  Our primary outcome for maternal depression using the MINI will be the proportion of women who meet MINI current MDD diagnostic criteria at 6 months.
Maternal Depressive Symptoms | 6 months
  Edinburgh Postnatal Depression Scale (EPDS): The EPDS is the 10-item gold standard measure of maternal depressive symptoms. A score >12 is consistent with PPD and changes in scores of 4 or more points are indicative of clinically significant improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van LIeshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh K, Layton H, Savoy CD, Ferro MA, Bieling PJ, Hicks A, Van Lieshout RJ. Online Public Health Nurse-Delivered Group Cognitive Behavioral Therapy for Postpartum Depression: A Randomized Controlled Trial During the COVID-19 Pandemic. J Clin Psychiatry. 2023 Jul 24;84(5):22m14726. doi: 10.4088/JCP.22m14726. PMID 37498661